CLINICAL TRIAL: NCT06506136
Title: Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial to Evaluate the Efficacy and Safety of Fluoxetine in Patients With Refractory Constipation Exhibiting Somatic Symptom Disorder Features
Brief Title: Evaluation of Fluoxetine for Refractory Constipation With Somatic Symptom Disorder Features
Acronym: REFLECT
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhifeng Zhao, PhD (Other)
Responsible Party: Sponsor-Investigator, Zhifeng Zhao, PhD, Dr., Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20242190
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Refractory Constipation; Somatic Symptom Disorder (DSM-5); Functional Constipation (FC)
Keywords: refractory constipation; fluoxetine; somatic symptom disorder; functional constipation
MeSH Terms: conditions — Constipation | interventions — Fluoxetine

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, double-blind, placebo-controlled "Parallel Assignment" design with two arms:
  Experimental Arm - Fluoxetine 20 mg qd
  Control Arm - Matching Placebo qd
  Participants are assigned in a 1 : 1 ratio by a central interactive web-response system, using permuted blocks stratified by study center and baseline CSBM frequency. Each participant receives only one intervention for the entire 12-week treatment period (plus taper/follow-up), with no crossover between arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluoxetine Treatment Group (Experimental)
  Interventions: Drug: Fluoxetine
- Placebo Control Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — Participants will receive fluoxetine tablets, 40 mg once daily, administered 30 minutes after breakfast for 12 weeks.
  Emergency Rescue Medications: For participants in both groups who cannot have a bowel movement for three consecutive days or have intolerable symptoms, the following rescue medications will be provided:
  polyethylene glycol：13.7 g enema Use of rescue medications must be recorded in the bowel movement diary and CRF, including date, time, and dosage. Rescue medications will be provided throughout the study but are not allowed within 48 hours before and after the first treatment. Distributed every two weeks, any bowel movements within 24 hours after rescue medication use will not count as CSBM.
  Arms: Fluoxetine Treatment Group
Drug: Placebo — Participants in the Placebo Control Group will receive placebo tablets that are identical in appearance and taste to the fluoxetine tablets. They will take one placebo tablet orally twice a day for 12 weeks, following the same schedule as the treatment group to maintain blinding.
  Emergency Rescue Medications: For participants in both groups who cannot have a bowel movement for three consecutive days or have intolerable symptoms, the following rescue medications will be provided:
  polyethylene glycol：13.7 g enema Use of rescue medications must be recorded in the bowel movement diary and CRF, including date, time, and dosage. Rescue medications will be provided throughout the study but are not allowed within 48 hours before and after the first treatment. Distributed every two weeks, any bowel movements within 24 hours after rescue medication use will not count as CSBM.
  Arms: Placebo Control Group

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled trial is to determine whether fluoxetine is effective and safe for adults with refractory constipation that exhibits Somatic Symptom Disorder (SSD) features-namely, persistent preoccupation with bowel function, heightened perception of defecatory discomfort, and clinically significant somatic symptom burden (PHQ-15 ≥ 10) in the absence of IBS-C abdominal pain criteria.

The study will address three primary questions:

Efficacy-Bowel Function:

• Does 12 weeks of fluoxetine increase Complete Spontaneous Bowel Movements (CSBM) and overall bowel-movement frequency compared with placebo?

Efficacy-Somatic Symptom Burden:

• Does fluoxetine reduce SSD severity, as measured by the Patient Health Questionnaire-15 (PHQ-15) and the Somatic Symptom Scale-8 (SSS-8)?

Safety and Tolerability:

• What adverse events occur during fluoxetine treatment, and how do their incidence and intensity compare with placebo?

ELIGIBILITY:
Participants in this study were recruited from a real-world outpatient constipation patient registry platform, which provides a comprehensive case database to support evidence-based research. Based on the characteristics of the primary target population identified in previous studies of fluoxetine, participants with refractory constipation were selected from the registry according to the following criteria:

All participants were required to meet the Rome IV diagnostic criteria for functional constipation.Specifically: 1) At least two of the following symptoms must be present during more than 25% of defecations: straining; lumpy or hard stools; sensation of incomplete evacuation; sensation of anorectal obstruction/blockage; manual maneuvers to facilitate defecation; fewer than three spontaneous bowel movements per week; 2) Loose stools are rarely present without the use of laxatives; 3) The criteria for IBS were not met.

Symptoms must have been present for at least six months prior to diagnosis, with the diagnostic criteria fulfilled during the last three months. Participants who met the diagnostic criteria were further assessed against the inclusion and exclusion criteria outlined below. Patients who did not meet any inclusion criteria or met any exclusion criteria were not recruited.

Inclusion criteria

1. Diagnosis of Functional Constipation (FC): Participants must meet the diagnostic criteria for functional constipation according to Rome IV criteria.
2. Low CSBM Frequency: During the 2-week screening period, participants must experience Complete Spontaneous Bowel Movements (CSBM) ≤ 2 times per week.
3. Unsatisfactory Previous Treatments: Participants must have been dissatisfied with previous treatments for functional constipation, having undergone at least 3 months of treatment, including laxatives or other prokinetic agents.
4. Diagnosis of Somatic Symptom Disorder (SSD): Participants must meet the diagnostic criteria for Somatic Symptom Disorder (SSD) according to DSM-5. All participants will undergo a semi-structured clinical interview based on DSM-5 criteria, conducted by professionals trained in SSD diagnosis.

   4.1. Criterion A: One or more physical symptoms that cause significant discomfort and/or disruption in daily life.

   4.2. Criterion B: At least one of the following: 1) Excessive and persistent thoughts about the severity of symptoms. 2) Persistent high anxiety about health or symptoms. 3) Excessive time and energy spent on health concerns or symptoms.

   4.3. Criterion C: The symptoms have persisted for at least 6 months.
5. Age Range: Participants must be between the ages of 18 and 60 years.
6. Not Participating in Other Ongoing Trials: Participants must not be involved in any other clinical trials during the study period.
7. Informed Consent: Participants must voluntarily agree to participate in the study and sign an informed consent form.

Exclusion criteria

1. Organic Diseases: Participants with organic diseases (e.g., tuberculosis, Crohn's disease, tumors, congenital megacolon), endocrine disorders (e.g., hypothyroidism), metabolic diseases (e.g., diabetes, thyroid dysfunction), or neurological disorders (e.g., Parkinson's disease).
2. Use of Medications Affecting Bowel Function: Participants who require long-term use of medications that may affect bowel function or induce constipation, such as Parkinson's medications, except for routine laxatives, antidiarrheal agents, and intestinal stimulants. Note: During the trial, participants are only allowed to use the specified emergency medications, and all medication use must be carefully recorded.
3. Chronic Pain or Substance Abuse: Participants with a history of chronic pain lasting more than 6 months or with a pain score ≥4 (based on the visual analog scale), or a history of substance abuse.
4. Mental Health Disorders: Participants diagnosed with psychiatric disorders before the study and continuously using psychiatric medications for more than 3 months, or those with a history of using psychiatric medications and/or corticosteroids for more than 3 months before the study.
5. Self-harm or Suicide Risk: Participants with a risk of self-harm or suicide, as assessed by a psychologist, or those requiring psychophysical interventions.
6. Allergic Reactions or Contraindications to Psychiatric Medications: Participants with a history of allergy to psychiatric medications, including fluoxetine, or those with liver or kidney dysfunction, or any contraindications for fluoxetine, such as prolonged QT interval on ECG.
7. Pregnant or Breastfeeding Women: Pregnant or breastfeeding women.
8. Other Malignant or Benign Tumors: Participants with other malignant or benign tumors or autoimmune diseases.
9. Chronic Diseases Impacting Life Quality: Participants with cardiovascular diseases, clotting disorders (e.g., those on long-term warfarin or heparin therapy), liver or kidney diseases, organ failure, cognitive disorders, aphasia, or any other chronic diseases requiring long-term medication, which may significantly affect their quality of life and the evaluation of treatment outcomes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy rate of fluoxetine treatment | Baseline (Week -2) through the end of Week 12 (treatment period)
  The primary efficacy endpoint is the proportion (%) of participants who achieve an increase of ≥ 1 complete spontaneous bowel movement (CSBM) per week relative to baseline in at least four of the twelve treatment weeks, a key indicator of therapeutic response in functional constipation (FC).

SECONDARY OUTCOMES:
Proportion of Participants Achieving ≥3 CSBM per Week | baseline and 12-week
  Percentage of participants who achieve at least 3 complete spontaneous bowel movements (CSBM) per week during the 12-week treatment period.
Change in the SBM compared to baseline over the 12-week treatment period | Baseline to Week-12
  Refers to a bowel movement occurring within the past 24 hours without the use of rescue medications or any other adjunctive methods (e.g., laxatives, enemas, suppositories, or digital maneuvers), including CSBM
Change from Baseline in Weekly CSBM Frequency | Baseline to Week-12
  The mean change in weekly complete spontaneous bowel movements (CSBM) compared to baseline.
Change in the average straining score for SBM over 12 weeks compared to baseline | Baseline to Week-12
  0 = no difficulty;
  1. = mild difficulty, straining required;
  2. = moderate difficulty, straining required;
  3. = severe difficulty, intense straining required.
Change in the abdominal bloating score compared to baseline over the 12-week treatment period | Baseline to Week-12
  Abdominal bloating will be assessed using a 5-point ordinal scale:
  1. = none;
  2. = mild;
  3. = moderate;
  4. = severe;
  5. = very severe.
Change in the average stool consistency score for SBM over 12 weeks compared to baseline | Baseline to Week-12
  Participants will self-report the stool consistency of each SBM using the Bristol Stool Form Scale
The change in KESS score from baseline to the end of the treatment period | Baseline to Week-12
  A validated questionnaire designed to quantify the severity and symptom profile of chronic constipation. It consists of 11 items, each scored from 0 to 4 based on symptom severity. Higher total scores indicate more severe constipation symptoms.
Change in PAC-QOL self-assessment scores from baseline | Baseline to Week-12
  A validated constipation-specific quality of life instrument developed to assess the impact of constipation on daily living. It includes 28 items covering four domains: physical discomfort, psychosocial discomfort, worries and concerns, and satisfaction, reflecting the effect of constipation over the past two weeks.
The change in GAD-7 score from baseline to the end of the treatment period | Baseline to Week-12
  Change in the Generalized Anxiety Disorder-7 (GAD-7) score from baseline to Week 12, assessing anxiety symptoms.
The change in PHQ-9 score from baseline to the end of the treatment period | Baseline to Week-12
  Change in the Patient Health Questionnaire-9 (PHQ-9) score from baseline to Week 12, assessing depressive symptoms.
The change in PHQ-15 score from baseline to the end of the treatment period | Baseline to Week-12
  Change in the Patient Health Questionnaire-15 (PHQ-15) score from baseline to Week 12, assessing somatic symptom severity related to SSD.
Incidence of adverse events | Weeks-2-12
  The proportion of participants experiencing adverse events in each treatment group during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Qingchuan Zhao, Prof., Study Chair — Xijing Hospital of Digestive Diseases
Locations (2):
- China (2):
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact zhaozhifeng@outlook.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: For more information or to submit a request, please contact zhaozhifeng@outlook.com.
URL: https://prsinfo.clinicaltrials.gov/definitions.html